CLINICAL TRIAL: NCT02548013
Title: Is Outpatient Management of PPROM Equivalent to Hospital Management
Brief Title: Preterm Premature Rupture of Membranes, Outpatient Management vs Inpatient Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, dina mostafa ibrahim, specialist, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ain Shams MS PPROM
Record Dates: First submitted 2015-08-25; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Preterm Premature Rupture of Membranes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home management (Experimental): outpatient management patients if stable will be discharged to continue treatment at home
  Interventions: Other: outpatient management
- hospital management (Active Comparator): Inpatient management patients will continue there treatment in hospital till delivery
  Interventions: Other: Inpatient management

INTERVENTIONS:
Other: outpatient management — patients if stable will be discharged to continue treatment at home
  Arms: Home management
Other: Inpatient management — patients will continue there treatment in hospital till delivery
  Arms: hospital management

SUMMARY:
This study is to compare the maternal and neonatal outcomes in the patients with PPROM who are managed at home versus those managed at hospital, half the patients will be managed at home and the other half will be managed inpatient.

DETAILED DESCRIPTION:
Now the current practice is to manage patients with PPROM at hospital, however it is not known yet whether this practice is better than outpatient management as regard maternal and neonatal outcome.

There is some recent evidence that home management of PPROM is safe for both mother and neonate, home management is also more convenient with less expenses.

ELIGIBILITY:
Inclusion Criteria:

1. PPROM with gestational age between 27 to 34 weeks
2. Cephalic presentation
3. Clear amniotic fluid
4. Oral temperature > 38 C
5. Near distance from the hospital (the patient can reach hospital within one hour )
6. Home environment safe and amenable to rest , availability of family support such as a sister or mother who will help the patient at home .
7. Maternal and fetal condition remain stable after hospitalization for 72 hours

Exclusion Criteria:

1. Patient with equivocal diagnosis of rupture of membranes
2. advanced labor
3. intrauterine infection
4. vaginal bleeding or
5. non reassuring fetal heart rate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 560 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
rate occurence of Neonatal sepsis | 48 hours after delivery
  proven neonatal infection with positive blood culture within 48 hours after birth, or culture proven neonatal pneumonia or meningitis

SECONDARY OUTCOMES:
rate of occurence of Maternal morbidity | 48 hours after delivery
  including chorioamnionitis , endometritis , septicaemia, admission to intensive care unit, organ failure, major postpartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Maged R Aboseda, professor, Study Chair — Ain Shams University maternity hospital
Locations (1):
- Ain Shams Maternity hospital, Cairo, Abbasya, Egypt